CLINICAL TRIAL: NCT02178995
Title: Methylphenidate Treatment of Attentional and Cognitive Deficits in Epilepsy
Brief Title: Methylphenidate Treatment of Attention Deficits in Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kimford Jay Meador (Other)
Responsible Party: Sponsor-Investigator, Kimford Jay Meador, Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MPH in epilepsy
Record Dates: First submitted 2014-06-24; First posted 2014-07-01 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Epilepsy; Cognitive Deficits; Attention Deficits
MeSH Terms: conditions — Epilepsy; Cognition Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Healthy Controls (No Intervention): Healthy controls completed the same neurocognitive batteries and neuropsychiatric questionnaires as individuals with epilepsy, but were not exposed to study medication.
  Healthy controls were included primarily for use in the open-label comparison. They did not receive blinded medication during the 'double-blind' portion and their data was not used in the 'double-blind' comparison. In order to control for test/re-test variables, they completed testing during the 'double-blind' portion, so that they completed testing an equivalent number of times to the epilepsy patients in the 'open-label' portion.
- Participants With Epilepsy (Open-label) (Experimental): Following the final randomized visit, interested participants were prescribed 10mg of methylphenidate twice daily, increased to 20mg of methylphenidate twice daily as tolerated. After a four week treatment trial, their scores on the batteries and questionnaires were again assessed.
  Interventions: Drug: Methylphenidate
- 10mg, 20mg, Then Placebo (Double-blind) (Experimental): Participants received three single doses in randomized order of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and completed cognitive testing and neuropsychiatric questionnaires. This single-dose phase was followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy first received blinded, single-dose capsules which contained either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate. At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
  Interventions: Drug: Methylphenidate
- 10mg, Placebo, Then 20mg (Double-blind) (Experimental): Participants received three single doses in randomized order of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and completed cognitive testing and neuropsychiatric questionnaires. This single-dose phase was followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy first received blinded, single-dose capsules which contained either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate. At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
  Interventions: Drug: Methylphenidate
- Placebo, 20mg, Then 10mg (Double-blind) (Experimental): Participants received three single doses in randomized order of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and completed cognitive testing and neuropsychiatric questionnaires. This single-dose phase was followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy first received blinded, single-dose capsules which contained either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate. At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
  Interventions: Drug: Methylphenidate
- Placebo, 10mg, Then 20mg (Double-blind) (Experimental): Participants received three single doses in randomized order of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and completed cognitive testing and neuropsychiatric questionnaires. This single-dose phase was followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy first received blinded, single-dose capsules which contained either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate. At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
  Interventions: Drug: Methylphenidate
- 20mg, Placebo, Then 10mg (Double-blind) (Experimental): Participants received three single doses in randomized order of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and completed cognitive testing and neuropsychiatric questionnaires. This single-dose phase was followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy first received blinded, single-dose capsules which contained either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate. At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
  Interventions: Drug: Methylphenidate
- 20mg, 10mg, Then Placebo - Double-blind (Experimental): Participants received three single doses in randomized order of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and completed cognitive testing and neuropsychiatric questionnaires. This single-dose phase was followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy first received blinded, single-dose capsules which contained either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate. At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
  Interventions: Drug: Methylphenidate
- 40mg, 20mg, Then Placebo (One Participant) (Experimental): This study was originally intended to use 40mg, 20mg, and placebo doses rather than 20mg, 10mg, and placebo. This individual developed tachycardia (see adverse events) on the 40mg dose, and was withdrawn from the double-blind portion as a result. We removed the 40mg doses from this study and replaced them with 10mg doses. No other participant received a 40mg dose. This participant rejoined the open-label portion after consultation with his PCP due to significant perceived benefit from the MPH dose.
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — Participants with epilepsy will first receive blinded, single-dose capsules which contain either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate.
  At each visit, they will receive one capsule and then complete the neurocognitive batteries and neuropsychiatric questionnaires. There will be no medication administered between visits during this time. Following the final randomized visit, interested participants will be prescribed 10mg of methylphenidate twice daily, to be increased to 20mg of methylphenidate twice daily. After four weeks, their scores on the batteries and questionnaires will again be assessed.
  Other Names: Ritalin
  Arms: 10mg, 20mg, Then Placebo (Double-blind); 10mg, Placebo, Then 20mg (Double-blind); 20mg, 10mg, Then Placebo - Double-blind; 20mg, Placebo, Then 10mg (Double-blind); 40mg, 20mg, Then Placebo (One Participant); Participants With Epilepsy (Open-label); Placebo, 10mg, Then 20mg (Double-blind); Placebo, 20mg, Then 10mg (Double-blind)

SUMMARY:
Methylphenidate (MPH) has long been used to improve attention and cognitive difficulties associated with ADHD, including in children with ADHD and epilepsy (Torres et al., 2008). Methylphenidate (MPH) is also helpful in treating attention and other cognitive difficulties in a variety of other neurological and medical conditions (Kajs-Wyllie, 2002; Prommer, 2012). We seek to evaluate the potential efficacy and safety of this medication in treating attention deficits, as well as other cognitive difficulties, experienced by adult patients with epilepsy.

To our knowledge, there are currently very few studies which explicitly examine the impact of MPH on measureable attention deficits and other cognitive deficits in adult patients with epilepsy. We hope to quantify what impact, if any, methylphenidate has on attention, in addition to other specific measureable cognitive functions, in patients with cognitive complaints and epilepsy, and contribute to a growing body of evidence which supports the safety of methylphenidate's use for attention deficits in patients with epilepsy. As other effective treatments for attention and other cognitive difficulties in patients with epilepsy are not currently available, MPH could represent an important option in the treatment of such patients.

DETAILED DESCRIPTION:
Prospective participants with seizures will be identified primarily through the Stanford Neurology and Neuropsychiatry clinics and Stanford Medical Center, with the assistance of clinic staff and providers. Participants may also be identified and referred by their physicians in the community as well. Informational fliers will be distributed to these clinics and throughout Stanford Medical Center and Stanford campus in order to identify participants with epilepsy as well as healthy volunteers. Prospective participants may also contact study staff directly via contact information listed on the flier or provided to them by their providers. Those identified will be contacted, either in person or by telephone, by study staff.

A telephone or in-person pre-screening will occur, expected to last approximately 20-30 minutes, in order to determine eligibility for the study, interest in participating, and any questions related to the study. A brief summary of study procedures and goals will be reviewed during this pre-screening. Participants who meet inclusion/exclusion criteria may take part in an initial in-person visit at Stanford Medical Center, where informed consent will be obtained and signed (see attached informed consent form). Any additional history needed in order to confirm a participant's eligibility will be reviewed at this visit. If the individual chooses to proceed, the participant's blood pressure and heartrate will be measured, and if necessary (because a recent physical exam including cardiac auscultation is not available), a brief physical exam will be performed by a licensed physician. If vital signs and exam (if necessary) are normal, participants will be asked to complete neuropsychiatric questionnaires, self-report questionnaires, a quality-of-life questionnaire, and a seizure diary. The full 40-minute neurocognitive battery will be performed, and baseline scores obtained.

Participants will be asked to complete the seizure diary once per week, either in-person at their visits or at home. Thereafter, the participant will be asked to attend at least three additional 2-hour sessions at Stanford Medical Center. The participant will be asked to avoid taking any non-routine sedating medications within 24 hours of his/her scheduled visit, and to refrain from eating, drinking caffeine, or smoking for 2 hours prior to his/her visit. When the participant arrives, they will be given either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate (randomized and blinded by the research pharmacy), and asked to remain within the hospital for 1 hour prior to testing to allow the medication to enter their system. Both study staff and the participant will be blinded to whether they are receiving active medication or placebo. During this time, the participant will complete self-report questionnaires reporting any medication changes, medical events, or significant adverse events, and their seizure diary will be reviewed and kept by study staff. After this, the full neurocognitive battery will be completed. Following the completion of neurocognitive testing, the participant's next visit will be scheduled for approximately the same time of day in approximately one week, and payment will be provided. This procedure will be repeated for the next two visits. Participants will not receive any additional study drug during this period other than the single dose they receive in-person.

At the participant's fourth visit, they will be asked to repeat the neuropsychiatric questionnaires from visit #1, as well as the usual self-report forms and seizure diary. Heartrate and blood pressure will be obtained again prior to the administration of the neurocognitive battery. At the end of the fourth visit, participants will be asked if they wish to take part in the four-week open-label phase of this study, designed to evaluate the ongoing efficacy and safety of methylphenidate for use in patients with epilepsy. Regardless of their answer, payment will be provided for their fourth visit.

Those participants who are interested in participating in the open-label trial will be provided with a prescription for two weeks of methylphenidate 10mg PO BID, followed by two weeks of methylphenidate 20mg PO BID. Participants will be provided with copies of the seizure diary and asked to complete it weekly. Participants will be able to contact the protocol director by phone to report any significant side effects or adverse events during this trial. At the protocol director's discretion, in keeping with standard of care for this medication, the dosage of the medication may be lowered (minimum dose 5mg PO BID) in response to any side effects experienced by participants during this period.

Participants in the open-label trial will be asked to return after four more weeks for a fifth and final visit. Participants will again be asked to refrain from eating, caffeine, and nicotine for 2 hours prior to their visit, and will take their prescribed methylphenidate upon arriving at Stanford Medical Center. Participants will wait 1 hour for the medication to enter their system, during which time they will complete neuropsychiatric and self-report questionnaires as before, their seizure diaries will be reviewed, and their heart rate and blood pressure will again be measured. The cognitive battery will be administered again. Afterwards, any participant questions will be answered and final financial compensation will be provided, and the participant's involvement has ended. Data will remain blinded until the completion of the study. Participants wishing to receive the active medication following the termination of the open-label phase of the study may do so at the discretion of their physicians.

ELIGIBILITY:
Inclusion Criteria:

1. For participants with seizures:

   * H/o seizures of any cause
   * Subjective cognitive complaints
   * Stable antiepileptic drug doses which are not expected to change during the study
   * Recent normal cardiac auscultation (may be done prior to enrollment by personal physician or study staff)
   * Neurologist's judgement that participant is clinically appropriate for this study
2. For healthy volunteers

   * No history of seizures or other neurological disorders
   * No history of cognitive complaints for any reason (including ADHD)
   * Not on any medications which would interfere w/ cognitive testing
3. English fluency

Exclusion Criteria:

1. IQ
2. History of an adverse reaction to methylphenidate
3. Age >65 or <18
4. Personal medical history of

   1. Arrhythmias,
   2. Structural cardiac disease,
   3. Other cardiac abnormality
   4. Uncontrolled hypertension (>150/95) during study. For those with BP >140/90 & <150/95, they will be monitored during the study and refer them for treatment if their BP remains elevated throughout the study.
   5. Uncontrolled tachycardia during study
   6. Progressive neurological disorders which may interfere w/ cognition for reasons other than seizures
   7. Glaucoma
   8. Other medical or neurological illnesses or symptoms which may interfere with cognition or medication (e.g., severe liver or renal disease, active infections, etc), or which make use of the medication inappropriate (e.g., severe agitation/anxiety).
   9. Intellectual disability sufficient to render a participant unable to consent
   10. Status epilepticus within the last year
   11. Neurosurgery which would be expected to interfere with study tasks within the last 6 months.
5. Substance use history

   1. Met criteria for substance use disorder within the past year
   2. Active illicit substance use
   3. Alcohol use meeting criteria for substance abuse
   4. Unwillingness to abstain from alcohol w/in 24 hours of testing
6. Personal psychiatric history

   1. History of a primary psychotic disorder, such as schizophrenia, or mania.
   2. History of suicide attempts within the last year
   3. Active suicidality
7. Severe cognitive impairments (e.g. aphasia) which render a participant unable to consent
8. Currently receiving medications which would be expected to interfere with the study tasks, if they cannot be held for study visits;
9. Pregnancy or active breastfeeding;
10. Women of childbearing potential who are sexually active and not willing or able to use a contraceptive strategy during the course of the study.
11. Any other factor which may interfere w/ a participant's ability to consent or to complete the required cognitive tasks, or may significantly interfere with their performance on the required tests
12. Concomitant use of an MAOI (if receiving methylphenidate during this study), or use of an MAOI within the last 14 days prior to receiving methylphenidate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse M Adams, MD, Study Director — Stanford University; Kimford Meador, MD, Principal Investigator — Stanford University; John Barry, MD, Study Chair — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Derived] Adams J, Alipio-Jocson V, Inoyama K, Bartlett V, Sandhu S, Oso J, Barry JJ, Loring DW, Meador K. Methylphenidate, cognition, and epilepsy: A double-blind, placebo-controlled, single-dose study. Neurology. 2017 Jan 31;88(5):470-476. doi: 10.1212/WNL.0000000000003564. Epub 2016 Dec 28. PMID 28031390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled primarily through the Stanford Neurology and Neuropsychiatry clinics between August 2014 and July 2015.
Pre-assignment Details: 4 participants signed their consent form, but did not complete any study visits and therefore produced no study data. Therefore, 55 participants are 'enrolled,' but only 51 actually participated in the study flow.
Groups:
- Placebo, 20mg, Then 10mg (Double-blind; Placebo, 10mg, Then 20mg (Double-blind); 20mg, Placebo, Then 10mg (Double-blind); 20mg, 10mg, Then Placebo - Double-blind: Participants received three single doses in randomized order of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and completed cognitive testing and neuropsychiatric questionnaires. This single-dose phase was followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy first received blinded, single-dose capsules which contained either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate.
  At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
Period: Double Blind
Arm/Group | Participants With Epilepsy (Open-label) | Healthy Controls | 10mg, 20mg, Then Placebo (Double-blind) | 10mg, Placebo, Then 20mg (Double-blind) | Placebo, 20mg, Then 10mg (Double-blind | Placebo, 10mg, Then 20mg (Double-blind) | 20mg, Placebo, Then 10mg (Double-blind) | 20mg, 10mg, Then Placebo - Double-blind | 40mg, 20mg, Then Placebo (One Participant)
Started | 0 | 16 | 5 | 6 | 6 | 6 | 5 | 6 | 1
Completed | 0 | 15 | 5 | 6 | 6 | 5 | 5 | 4 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Open Label
Arm/Group | Participants With Epilepsy (Open-label) | Healthy Controls | 10mg, 20mg, Then Placebo (Double-blind) | 10mg, Placebo, Then 20mg (Double-blind) | Placebo, 20mg, Then 10mg (Double-blind | Placebo, 10mg, Then 20mg (Double-blind) | 20mg, Placebo, Then 10mg (Double-blind) | 20mg, 10mg, Then Placebo - Double-blind | 40mg, 20mg, Then Placebo (One Participant)
Started | 30 (2 declined to join open-label. 1 withdrew from double-blind but rejoined open-label due to benefit.) | 14 (One was lost to follow-up after completion of visit 4.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 28 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total number of individuals who signed consents = 55. 4 of these individuals with epilepsy signed their consent but did not follow through and participate in the study. The remaining 51 (35 epilepsy, 16 controls) are represented here.
Groups:
- Participants With Epilepsy: Participants received three single doses of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and completed cognitive testing and neuropsychiatric questionnaires. This single-dose phase was followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy first received blinded, single-dose capsules which contained either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate.
  At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time. Following the final randomized visit, interested participants were prescribed 10mg of methylphenidate twice daily, increased to 20mg of methylphenidate twice daily as tolerated. After four weeks, their scores on the batteries and questionnaires were again assessed.
- Healthy Controls: Healthy controls completed the same neurocognitive batteries and neuropsychiatric questionnaires as individuals with epilepsy, but were not exposed to study medication.
- Total: Total of all reporting groups
Arm/Group | Participants With Epilepsy | Healthy Controls | Total
Number analyzed (Participants) | 35 | 16 | 51
Age, Continuous [Mean (Full Range); unit: years] | 37 [20 to 64] | 45 [22 to 62] | 39.5 [20 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 16 | 6 | 22
Mean years of education [Mean (Full Range); unit: years] | 15 [12 to 20] | 15 [12 to 18] | 15 [12 to 20]
Mean duration of epilepsy [Mean (Full Range); unit: years] | 12.5 [1 to 41] | 0 [0 to 0] | NA [NA to NA] — Healthy controls do not have epilepsy.
Seizure type [Number; unit: participants]
  Focal | 26 | 0 | 26
  Generalized | 6 | 0 | 6
  Unclassified (GTCS) | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Conners' Continuous Performance Test (CPT) (Double-blind Portion, Primary Variables)
Description: Scores on this test measure attentiveness/vigilance and response time. Primary measures are: D', HRTSD D' represents 'detectability,' and is a derived statistic which measures a participant's ability to distinguish target stimuli from non-target stimuli, and incorporates response time and accuracy factors. The equation for deriving it is proprietary to the test which markets the CPT. A higher, or less negative, score is considered WORSE.
  HRTSD represents the standard deviation of participant hit reaction time data, as measured for a variety of different stimuli types across the trial. It is a measure of the participant's ability to maintain attention across the trial. A higher score represents more variability and is considered WORSE.
Time Frame: difference in scores on specific variables between MPH 20mg, 10mg, and placebo (randomized to administration at weeks 2, 3, or 4)
Measure: Mean (Standard Deviation); unit: Units
Groups:
- Participants With Epilepsy: Placebo: Methylphenidate: Participants received blinded, single-dose capsules during either visit 2, 3, or 4. During one of these visits, they received the placebo capsule.
  At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
- Participants With Epilepsy: Methylphenidate 10 mg Dose: Participants received blinded, single-dose capsules of during visits 2, 3, and 4. During one of these visits, they received the methylphenidate 10 mg dose.
  At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
- Participants With Epilepsy: Methylphenidate 20 mg: Participants received blinded, single-dose capsules of during visits 2, 3, and 4. During one of these visits, they received the methylphenidate 20 mg dose.
  At each visit, they received one capsule and then completed the neurocognitive batteries and neuropsychiatric questionnaires. There was no medication administered between visits during this time.
Arm/Group | Participants With Epilepsy: Placebo | Participants With Epilepsy: Methylphenidate 10 mg Dose | Participants With Epilepsy: Methylphenidate 20 mg
Number analyzed (Participants) | 31 | 31 | 31
Units
  D' | -3.3 (0.9) | -3.58 (0.78) | -3.66 (0.77)
  HRTSD | 0.19 (0.048) | 0.17 (0.034) | 0.17 (0.036)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Test type: Superiority or Other; p = 0.037, ANOVA — HRTSD p-value = 0.037; p < 0.05 considered significant; Within-subjects contrasts, n=31, df=1
Statistical Analysis 2: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Test type: Superiority or Other; p = 0.055, ANOVA — D' p = 0.055. p < 0.05 considered significant; Within-subjects contrasts, placebo v 10mg v 20mg
Statistical Analysis 3: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; HRTSD 10mg vs 20mg; Test type: Superiority or Other; p = 0.758, t-test, 2 sided
Statistical Analysis 4: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; d' 10mg vs 20mg; Test type: Superiority or Other; p = 0.499, t-test, 2 sided

2. Primary Outcome: Symbol-digit Matching Test (Double-blind Portion)
Description: Symbol-digit matching test is a measure processing speed and working memory. The task involves matching nonsense symbols with numbers based on a key as quickly as possible within 90s. Score represents the number of correct responses within the time frame. Minimum score is 0. There is not a meaningful 'maximum' score, as there are too many symbols for a participant to successfully complete within the allotted time. A higher score is better.
Time Frame: Difference in scores between MPH 20mg, 10mg, or placebo during double-blind portion during which medication was randomized to weeks 2, 3, or 4.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Participants With Epilepsy: Placebo | Participants With Epilepsy: Methylphenidate 10 mg Dose | Participants With Epilepsy: Methylphenidate 20 mg
Number analyzed (Participants) | 31 | 31 | 31
points | 49.8 (11.9) | 52.2 (11.6) | 50.6 (11.3)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Test type: Superiority or Other; p = 0.008, ANOVA
Statistical Analysis 2: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; SDMT 10mg vs 20mg; Test type: Superiority or Other; p = 0.071, t-test, 2 sided

3. Primary Outcome: MCG Paragraph Memory Test (Double-blind Portion)
Description: MCG paragraph memory test is a measure of verbal memory. Participants are read aloud a long, detailed story, and are then asked to immediately repeat all information they can remember from the story. Each pertinent story element (as pre-defined on a key) is considered 1 correct response. Minimum score is 0, maximum is 100. A higher score is better.
Time Frame: Difference in scores between MPH 20mg, 10mg, or placebo, randomized to be given at weeks 2, 3, or 4
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Participants With Epilepsy: Placebo | Participants With Epilepsy: Methylphenidate 10 mg Dose | Participants With Epilepsy: Methylphenidate 20 mg
Number analyzed (Participants) | 31 | 31 | 31
Points | 25.2 (14.8) | 27.4 (15.4) | 28 (15.3)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Test type: Superiority or Other; p = 0.154, ANOVA
Statistical Analysis 2: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; MCG 10mg vs 20mg; Test type: Superiority or Other; p = 0.779, t-test, 2 sided

4. Primary Outcome: Conners CPT Outcomes (Primary Variables) (Open-Label Portion)
Description: Within-groups comparison (between visit 1 and visit 5 within patients with epilepsy, comparing scores at baseline to scores on methylphenidate) as well as a comparison against healthy controls who repeated the cognitive measures an equal number of times (to assess and control for test/retest and placebo improvements).
  D' represents 'detectability,' and is a derived statistic which measures a participant's ability to distinguish target stimuli from non-target stimuli, and incorporates response time and accuracy factors. The equation for deriving it is proprietary to the test which markets the CPT. A higher, or less negative, score is considered WORSE.
  HRTSD represents the standard deviation of participant hit reaction time data, as measured for a variety of different stimuli types across the trial. It is a measure of the participant's ability to maintain attention across the trial. A higher score represents more variability and is considered WORSE.
Time Frame: Difference between scores at baseline (visit 1) and on methylphenidate open-label (visit 5), compared to untreated healthy controls
Population: PLEASE NOTE: One participant with epilepsy did not record any usable data for Conners CPT due to pressing the wrong key throughout large portions of the trial. Therefore, he is not included in CPT variables (but is included in other analyses).
Measure: Mean (Standard Deviation); unit: Units
Groups:
- Participants With Epilepsy: Visit 1 (Baseline): At visit 1, participants underwent neurocognitive batteries and neuropsychiatric questionnaires for baseline assessment. No medications were given at this visit.
- Participants With Epilepsy: Visit 5 (Open Label): Following the final randomized visit, interested participants were prescribed 10mg of methylphenidate twice daily, increased to 20mg of methylphenidate twice daily as tolerated. After four weeks, their scores on the batteries and questionnaires were again assessed.
- Healthy Controls: Visit 1 (Baseline); Healthy Controls: Visit 5: Healthy controls completed the same neurocognitive batteries and neuropsychiatric questionnaires as individuals with epilepsy, but were not exposed to study medication.
  Healthy controls were included primarily for use in the open-label comparison. They did not receive blinded medication during the 'double-blind' portion and their data was not used in the 'double-blind' comparison. In order to control for test/re-test variables, they completed testing during the 'double-blind' portion, so that they completed testing an equivalent number of times to the epilepsy patients in the 'open-label' portion.
Arm/Group | Participants With Epilepsy: Visit 1 (Baseline) | Participants With Epilepsy: Visit 5 (Open Label) | Healthy Controls: Visit 1 (Baseline) | Healthy Controls: Visit 5
Number analyzed (Participants) | 27 | 27 | 14 | 14
Units
  HRTSD | 0.22 (0.04) | 0.16 (0.03) | 0.20 (0.04) | 0.15 (0.03)
  D' | -2.9 (0.9) | -3.8 (0.7) | -3.7 (0.5) | -4.2 (0.8)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); Intra-group comparison, HRTSD; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — HRTSD P<0.0001
Statistical Analysis 2: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Intra-group comparison, HRTSD, healthy controls; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — HRTSD p <0.001 for healthy controls
Statistical Analysis 3: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Between-group comparisons by 2-way ANOVA, HRTSD; Test type: Superiority or Other; p = 0.322, ANOVA
Statistical Analysis 4: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); Intra-group comparison, epilepsy, D'; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Intra-group analysis, healthy controls, d'; Test type: Superiority or Other; p = 0.037, t-test, 2 sided
Statistical Analysis 6: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Intra-group analysis by 2-way ANOVA, d'; Test type: Superiority or Other; p = 0.08, ANOVA

5. Primary Outcome: Symbol-digit Matching Test (Open Label Phase)
Description: as for outcome 2
Time Frame: The single-dose double blind phase was followed by an open-label 4-week treatment phase.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Participants With Epilepsy: Visit 1 (Baseline) | Participants With Epilepsy: Visit 5 (Open Label) | Healthy Controls: Visit 1 (Baseline) | Healthy Controls: Visit 5
Number analyzed (Participants) | 28 | 28 | 14 | 14
points | 48.1 (11.6) | 53.8 (12.0) | 55.9 (9.2) | 60.1 (8.9)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); Test type: Superiority or Other; p = 0.003, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Test type: Superiority or Other; p = 0.022, t-test, 2 sided
Statistical Analysis 3: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Group x time interaction by 2-way ANOVA; Test type: Superiority or Other; p = 0.443, ANOVA

6. Primary Outcome: MCG (Open-label Portion)
Description: MCG paragraph memory test is a measure verbal memory. Participants are read aloud a long, detailed story, and are then asked to immediately repeat all information they can remember from the story. Each pertinent story element (as pre-defined on a key) is considered 1 correct response. Minimum score is 0, maximum is 100. A higher score is better.
Time Frame: The single-dose double blind phase was followed by an open-label 4-week treatment phase.
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Participants With Epilepsy: Visit 1 (Baseline) | Participants With Epilepsy: Visit 5 (Open Label) | Healthy Controls: Visit 1 (Baseline) | Healthy Controls: Visit 5
Number analyzed (Participants) | 28 | 28 | 14 | 14
Points | 18.6 (13.4) | 30.5 (14.7) | 32.7 (16.3) | 44.9 (19.6)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Test type: Superiority or Other; p = 0.004, t-test, 2 sided
Statistical Analysis 3: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Between-groups analysis by 2-way ANOVA; Test type: Superiority or Other; p = 0.906, ANOVA

7. Primary Outcome: Seizure Frequency (Open-label Portion)
Description: Seizures per 28 'at-risk' days. This is a comparison of 28 days prior to baseline visit as compared to seizure rate while taking methylphenidate, adjusted to provide a 'number of seizures per 28 days' measurement.
Time Frame: Randomized portion is followed by 1-month open-label portion.
Population: This analysis only compares the 28 participants who were present in both groups. Participants who participated only in the double-blind portion are represented in that analysis.
Measure: Mean (Standard Deviation); unit: Seizures per 28 at-risk days
Groups:
- Participants With Epilepsy (Baseline): Participants will receive three single doses of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and will complete cognitive testing and neuropsychiatric questionnaires. This single-dose phase will be followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy will first receive blinded, single-dose capsules which contain either:
  Placebo 20mg of methylphenidate or 10mg of methylphenidate.
  At each visit, they will receive one capsule and then complete the neurocognitive batteries and neuropsychiatric questionnaires. There will be no medication administered between visits during this time. Following the final randomized visit, interested participants will be prescribed 10mg of methylphenidate twice daily, to be increased to 20mg of methylphenidate twice daily. After four weeks, their scores on the batteries and questionnaires will again be assessed.
Arm/Group | Participants With Epilepsy (Baseline) | Participants With Epilepsy (Open-label Portion)
Number analyzed (Participants) | 28 | 28
Seizures per 28 at-risk days | 2.8 (6.2) | 2.4 (5.7)
Statistical Analysis 1: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Test type: Superiority or Other; p = 0.274, t-test, 2 sided

8. Primary Outcome: QOLIE-89 Aggregate Score
Description: QOLIE-89 is a questionnaire to assess quality of life and subjective cognitive effects. The aggregate score is the overall calculated score. Note: most of its questions are specific to patients with epilepsy, and therefore the questionnaire cannot be validly completed by healthy controls. Therefore, only participants with epilepsy completed the questionnaire.
  QOLIE aggregate scores and subscale scores are calculated based on individual patient responses throughout the survey, and according to scoring rules as determined by the creator of the questionnaire. Scores are rated 0 (worst) to 100 (best).
Time Frame: Change from baseline to end of methylphenidate open label treatment (end month 2)
Measure: Mean (Standard Deviation); unit: Points
Groups:
- Participants With Epilepsy (Open-label Portion): Note: Because the QOLIE-89 is specific to epilepsy populations, most of its questions are not applicable to healthy controls, and therefore healthy controls did not complete the QOLIE-89.
Arm/Group | Participants With Epilepsy (Baseline) | Participants With Epilepsy (Open-label Portion)
Number analyzed (Participants) | 28 | 28
Points | 60.2 (17.1) | 72.0 (16.2)
Statistical Analysis 1: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

9. Secondary Outcome: CPT Scores (Double-blind Portion) (Secondary Variables)
Description: Secondary variables in CPT: hits, omissions, commissions
  "Hits" represents the raw number of accurate responses to target stimuli, out of a maximum of 288. A higher number is better.
  "Omissions" are errors committed when a target stimuli is not appropriately responded to. A higher number is worse. Theoretically, the maximum number of omissions would be 288. A lower number is BETTER.
  "Commissions" are errors committed when a participant responds to a non-target stimuli. Because a participant may make multiple such errors for a given stimuli, there is no raw maximum. A lower number is BETTER.
Time Frame: Difference between scores on MPH 20mg, 10mg, or placebo during randomized visits weeks 2, 3, or 4
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Participants With Epilepsy: Placebo | Participants With Epilepsy: Methylphenidate 10 mg Dose | Participants With Epilepsy: Methylphenidate 20 mg
Number analyzed (Participants) | 31 | 31 | 31
Units
  Hits | 285.3 (4.5) | 286.9 (1.6) | 287 (2.7)
  Omissions | 0.9 (1.5) | 0.3 (0.4) | 0.3 (0.8)
  Commissions | 24 (19.9) | 21.5 (18.2) | 21.2 (15.1)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Test type: Superiority or Other; p = 0.04, ANOVA — Hits p = 0.04
Statistical Analysis 2: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Test type: Superiority or Other; p = 0.038, ANOVA — Omissions p = 0.038
Statistical Analysis 3: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Test type: Superiority or Other; p = 0.329, ANOVA — Commissions p = 0.329
Statistical Analysis 4: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Hits 10mg vs 20mg; Test type: Superiority or Other; p = 0.876, t-test, 2 sided
Statistical Analysis 5: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Omissions 10mg vs 20mg; Test type: Superiority or Other; p = 0.932, t-test, 2 sided
Statistical Analysis 6: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Commissions 10mg vs 20mg; Test type: Superiority or Other; p = 0.898, t-test, 2 sided

10. Secondary Outcome: Seizure Frequency/Severity (Double-blind Portion)
Description: as for outcome 7
Time Frame: Seizure rate during 28 days prior to study compared to during randomized, single-dose portion, rate adjusted to seizures per 28 patient days.
Population: Only participants who were present in both groups are included here.
Measure: Mean (Standard Deviation); unit: Seizures per 28 at-risk days
Arm/Group | Participants With Epilepsy (Baseline) | Participants With Epilepsy (Double-blind Portion)
Number analyzed (Participants) | 31 | 31
Seizures per 28 at-risk days | 2.5 (5.9) | 2.0 (5.5)
Statistical Analysis 1: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Double-blind Portion); Comparison of baseline rate of seizures (expressed as seizures per 28 days) pre-trial against the rate experienced during the double-blind portion of our trial; Test type: Superiority or Other; p = 0.7116, t-test, 2 sided

11. Secondary Outcome: QOLIE-89 Selected Cognitive Subscales (Open-label)
Description: Pre-selected secondary variables were cognitive subscales on the QOLIE-89 felt likely to be affected by MPH: attention/concentration; memory; language; energy/fatigue.
  QOLIE aggregate scores and subscale scores are calculated based on individual patient responses throughout the survey, and according to scoring rules as determined by the creator of the questionnaire. Scores are rated 0 (worst) to 100 (best).
Time Frame: Comparing baseline (visit 1) to end of open-label (end of week 8)
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Participants With Epilepsy (Baseline) | Participants With Epilepsy (Open-label Portion)
Number analyzed (Participants) | 28 | 28
Points
  Attention/Concentration | 50.4 (21.4) | 74.8 (19.5)
  Memory | 36.8 (27.0) | 59.7 (26.3)
  Language | 58.1 (27.0) | 72.3 (21.9)
  Energy/Fatigue | 45.9 (21.2) | 61.6 (19.4)
Statistical Analysis 1: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Attention/Concentration subscale; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Memory subscale; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Language subscale; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 4: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Energy/fatigue subscale; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

12. Secondary Outcome: CPT Outcomes (Secondary Variables) (Open-label Portion)
Description: Omissions, commissions, and hits
  "Hits" represents the raw number of accurate responses to target stimuli, out of a maximum of 288. A higher number is better.
  "Omissions" are errors committed when a target stimuli is not appropriately responded to. A higher number is worse. Theoretically, the maximum number of omissions would be 288. A lower number is BETTER.
  "Commissions" are errors committed when a participant responds to a non-target stimuli. Because a participant may make multiple such errors for a given stimuli, there is no raw maximum. A lower number is BETTER.
Time Frame: Baseline (Visit 1) vs end of Open-label (week 8)
Population: Note: one epilepsy participant's CPT data was invalid/unusable due to pressing the wrong button during the trial.
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Participants With Epilepsy: Visit 1 (Baseline) | Participants With Epilepsy: Visit 5 (Open Label) | Healthy Controls: Visit 1 (Baseline) | Healthy Controls: Visit 5
Number analyzed (Participants) | 27 | 27 | 14 | 14
Points
  Hits | 284.6 (5.1) | 287.6 (0.9) | 287 (1.2) | 287.6 (0.7)
  Omissions | 1.0 (1.4) | 0.1 (0.3) | 0.3 (0.3) | 0.1 (0.2)
  Commissions | 34.8 (18.4) | 18.5 (17.8) | 16.7 (9.7) | 13.2 (16.1)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); Hits v1 vs v5 epilepsy; Test type: Superiority or Other; p = 0.003, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Hits v1 vs v5 healthy; Test type: Superiority or Other; p = 0.033, t-test, 2 sided
Statistical Analysis 3: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; 2-way ANOVA epilepsy vs healthy hits; Test type: Superiority or Other; p = 0.079, ANOVA
Statistical Analysis 4: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); Omissions epilepsy v1 vs v5; Test type: Superiority or Other; p = 0.001, t-test, 2 sided
Statistical Analysis 5: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Omissions v1 vs v5 healthy; Test type: Superiority or Other; p = 0.029, t-test, 2 sided
Statistical Analysis 6: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Epilepsy v healthy ANOVA Omissions; Test type: Superiority or Other; p = 0.048, t-test, 2 sided
Statistical Analysis 7: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); Commissions v1 vs v5 epilepsy; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Commissions v1 vs v5 healthy; Test type: Superiority or Other; p = 0.42, t-test, 2 sided
Statistical Analysis 9: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Healthy vs epilepsy ANOVA (2-way) commissions; Test type: Superiority or Other; p = 0.019, ANOVA

13. Other Pre Specified Outcome: Adverse Events Profile (Open-Label)
Description: This is a side-effects reporting scale for anti-epileptic medications. Because it encompasses cognitive and non-cognitive side effects, it was not considered one of our main cognitive/quality of life outcomes of interest. It is used in other studies of AED side effects, however, so was included.
  The scale consists of 19 symptoms rated 1 (Never a problem) to 4 (Always or often a problem). Minimum score is 19, maximum score is 76. A higher score is WORSE.
Time Frame: Baseline (Visit 1) vs end of Open-label (week 8)
Measure: Mean (Standard Deviation); unit: Points
Groups:
- Participants With Epilepsy (Open-label Portion): Note: Because the questionnaire is specific to epilepsy populations, and the side-effects to AEDs, healthy controls did not complete the QOLIE-89.
Arm/Group | Participants With Epilepsy (Baseline) | Participants With Epilepsy (Open-label Portion)
Number analyzed (Participants) | 28 | 28
Points | 41.9 (8.5) | 34.4 (9.6)
Statistical Analysis 1: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

14. Other Pre Specified Outcome: Stimulant Side-effects Checklist
Description: This is a questionnaire covering common stimulant side-effects, intended to help monitor for any significant or common adverse effects.
  The scale lists 16 common stimulant side effects rated 0 (absent) to 9 (serious). Minimum score is 0, maximum is 144. A higher score is WORSE.
Time Frame: Baseline (Visit 1) vs end of Open-label (week 8)
Measure: Mean (Standard Deviation); unit: Points
Groups:
- Participants With Epilepsy (Open-label Portion): Note: Because the SSC is specific to medication side effects, healthy controls did not complete the questionnaire.
Arm/Group | Participants With Epilepsy (Baseline) | Participants With Epilepsy (Open-label Portion)
Number analyzed (Participants) | 28 | 28
Points | 37.2 (21.0) | 27.3 (23.1)
Statistical Analysis 1: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Test type: Superiority or Other; p = 0.003, t-test, 2 sided — Note: Stimulant side-effect score *decreased* with addition of open-label stimulant

15. Other Pre Specified Outcome: Neuropsychiatric Questionnaires
Description: Beck Depression Inventory, Beck Anxiety Inventory, Apathy Evaluation Scale. These were not primary or secondary variables of interest given methylphenidate's primary expected action being on cognition. Included given one author's interest, as other studies suggesting psychiatric improvements (particularly apathy and depression) with methylphenidate.
  BDI is a common clinical and research measure of depression. It has 21 questions and is scored 0 (no depression) to 63 (most severe depression). A higher score is worse.
  BAI is a measure of anxiety, which also has 21 questions and is scored 0 (no anxiety) to 63 (most severe anxiety). A higher score is worse.
  AES is a measure of clinical apathy, and is an 18-item scale. It rates symptoms as "not at all," "slightly," "somewhat," or "a lot," which are then converted to numerical values 1 (least apathy) to 4 (most apathy). Scores range from 18 (no apathy) to 72 (most apathy).
Time Frame: Baseline (Visit 1) vs end of Open-label (week 8)
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Participants With Epilepsy: Visit 1 (Baseline) | Participants With Epilepsy: Visit 5 (Open Label) | Healthy Controls: Visit 1 (Baseline) | Healthy Controls: Visit 5
Number analyzed (Participants) | 28 | 28 | 14 | 14
Points
  BDI | 9.6 (7.3) | 6.4 (6.1) | 2.0 (1.7) | 1.1 (1.5)
  BAI | 10.9 (11.1) | 9.6 (9.2) | 2.4 (5.1) | 1.7 (2.1)
  AES | 31.2 (5.6) | 28.7 (7.0) | 23.3 (5.0) | 22.9 (4.7)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); BDI epilepsy v1 vs v5; Test type: Superiority or Other; p = 0.014, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Healthy controls BDI v1 vs v5; Test type: Superiority or Other; p = 0.04, t-test, 2 sided
Statistical Analysis 3: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Between-group comparison 2-way ANOVA BDI; Test type: Superiority or Other; p = 0.191, t-test, 2 sided
Statistical Analysis 4: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); BAI visit 1 vs visit 5 epilepsy; Test type: Superiority or Other; p = 0.42, t-test, 2 sided
Statistical Analysis 5: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; BAI visit 1 vs visit 5 healthy controls; Test type: Superiority or Other; p = 0.477, t-test, 2 sided
Statistical Analysis 6: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Between-groups comparison 2-way ANOVA BAI; Test type: Superiority or Other; p = 0.792, ANOVA
Statistical Analysis 7: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); AES visit 1 vs visit 5 epilepsy; Test type: Superiority or Other; p = 0.045, t-test, 2 sided
Statistical Analysis 8: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; AES visit 1 vs visit 5 healthy controls; Test type: Superiority or Other; p = 0.646, t-test, 2 sided
Statistical Analysis 9: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Between-groups comparison 2-way ANOVA AES; Test type: Superiority or Other; p = 0.222, ANOVA

16. Post Hoc Outcome: QOLIE-89 Additional Subscales (Open-label)
Description: These are the remaining subscales of the QOLIE-89. These were not pre-specified variables of interest or intentional post-hoc analyses, but are automatically calculated in scoring the QOLIE-89 and are included ONLY for completeness of data submission.
  QOLIE aggregate scores and subscale scores are calculated based on individual patient responses throughout the survey, and according to scoring rules as determined by the creator of the questionnaire. Scores are rated 0 (worst) to 100 (best).
Time Frame: Visit 1 (baseline) vs end of open-label (week 8)
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Participants With Epilepsy (Baseline) | Participants With Epilepsy (Open-label Portion)
Number analyzed (Participants) | 28 | 28
Points
  Health Perceptions | 55.2 (21.4) | 63.4 (22.4)
  Overall QOL (pt rating) | 65.5 (18.4) | 73.0 (14.3)
  Physical Function | 78.0 (27.4) | 83.2 (22.4)
  Role Limitations (Emotional) | 67.8 (43.0) | 79.3 (30.0)
  Role Limitations (Physical) | 62.8 (36.4) | 82.8 (30.6)
  Pain | 70.4 (30.9) | 78.1 (22.8)
  Work/Driving/Social | 61.1 (27.0) | 69.5 (22.4)
  Emotional Wellbeing | 70.3 (17.0) | 75.1 (17.8)
  Health Discouragement | 66.4 (30.8) | 81.8 (21.3)
  Seizure Worry | 55.5 (28.9) | 61.9 (31.7)
  Medication Effects | 48.1 (28.7) | 50.9 (30.9)
  Social Support | 71.2 (23.4) | 73.0 (24.5)
  Social Isolation | 74.6 (27.6) | 81.4 (21.4)
Statistical Analysis 1: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Health Perceptions; Test type: Superiority or Other; p = 0.011, t-test, 2 sided
Statistical Analysis 2: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Overall QOL (subjectively rated by participants on the scale); Test type: Superiority or Other; p = 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Physical Function; Test type: Superiority or Other; p = 0.164, t-test, 2 sided
Statistical Analysis 4: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Role Limitations (Emotional); Test type: Superiority or Other; p = 0.065, t-test, 2 sided
Statistical Analysis 5: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Role Limitations (Physical); Test type: Superiority or Other; p = 0.014, t-test, 2 sided
Statistical Analysis 6: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Pain; Test type: Superiority or Other; p = 0.128, t-test, 2 sided
Statistical Analysis 7: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Work/Driving/Social; Test type: Superiority or Other; p = 0.026, t-test, 2 sided
Statistical Analysis 8: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Emotional Wellbeing; Test type: Superiority or Other; p = 0.077, t-test, 2 sided
Statistical Analysis 9: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Health Discouragement; Test type: Superiority or Other; p = 0.007, t-test, 2 sided
Statistical Analysis 10: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Seizure Worry; Test type: Superiority or Other; p = 0.063, t-test, 2 sided
Statistical Analysis 11: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Medication Effects; Test type: Superiority or Other; p = 0.609, t-test, 2 sided
Statistical Analysis 12: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Social Support; Test type: Superiority or Other; p = 0.626, t-test, 2 sided
Statistical Analysis 13: Comparison: Participants With Epilepsy (Baseline) vs Participants With Epilepsy (Open-label Portion); Social Isolation; Test type: Superiority or Other; p = 0.103, t-test, 2 sided

17. Post Hoc Outcome: Remaining CPT Variables (Open-label)
Description: These are automatically-calculated CPT variables which were not pre-specified variables of interest or intentional post-hoc analyses. They are included ONLY for completeness of data. They include hit reaction time (HRT), variability (VAR), and perseverations (PRS).
  Hit reaction time represents to the average number of milliseconds required for a participant to respond to target stimuli. There are no meaningful absolute minimum or maximum scores, though 101ms is the current fastest verified response time per our review. A higher score is WORSE.
  Variability refers to variations in response time across individual blocks of time within the trial. It differs from HRTSD in that HRTSD measures variability across the entire trial. Minimum is 0. There are no absolute maximums. A higher score is WORSE.
  Perseverations are errors made either faster than physiologically possible (<100ms). Minimum is 0, there is no maximum. Higher scores are WORSE.
Time Frame: Baseline vs end of open-label (week 8)
Population: Note: One participant's CPT data was invalid
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Participants With Epilepsy: Visit 1 (Baseline) | Participants With Epilepsy: Visit 5 (Open Label) | Healthy Controls: Visit 1 (Baseline) | Healthy Controls: Visit 5
Number analyzed (Participants) | 27 | 27 | 14 | 14
Units
  Variability (units) | 0.05 (0.02) | 0.04 (0.008) | 0.042 (0.01) | 0.035 (0.009)
  Perseverations (units) | 0.2 (0.5) | 0.01 (0.05) | 0.08 (0.2) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); Variability v1 vs v5 epilepsy; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Variability v1 vs v5 healthy; Test type: Superiority or Other; p = 0.096, t-test, 2 sided
Statistical Analysis 3: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Variability 2-way ANOVA healthy vs epilepsy; Test type: Superiority or Other; p = 0.136, ANOVA
Statistical Analysis 4: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); Perseverations v1 vs v5 epilepsy; Test type: Superiority or Other; p = 0.17, t-test, 2 sided
Statistical Analysis 5: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Perseverations v1 vs v5 healthy; Test type: Superiority or Other; p = 0.104, t-test, 2 sided
Statistical Analysis 6: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; Perseverations 2-way ANOVA healthy vs epilepsy; Test type: Superiority or Other; p = 0.661, ANOVA

18. Post Hoc Outcome: Remaining CPT Variables (Double-blind Portion)
Description: Remaining CPT variables are automatically calculated by the program. They were not pre-specified variables of interest nor intentional post-hoc analyses. They are included ONLY for completeness of data submission.
  Hit reaction time represents to the average number of milliseconds required for a participant to respond to target stimuli. There are no meaningful absolute minimum or maximum scores, though 101ms is the current fastest verified response time per our review. A higher score is WORSE.
  Variability refers to variations in response time across individual blocks of time within the trial. It differs from HRTSD in that HRTSD measures variability across the entire trial. Minimum is 0. There are no absolute maximums. A higher score is WORSE.
  Perseverations are errors made either faster than physiologically possible (<100ms). Minimum is 0, there is no maximum. Higher scores are WORSE.
Time Frame: Placebo vs 10mg vs 20mg (visits 2, 3, 4)
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Participants With Epilepsy: Placebo | Participants With Epilepsy: Methylphenidate 10 mg Dose | Participants With Epilepsy: Methylphenidate 20 mg
Number analyzed (Participants) | 31 | 31 | 31
Units
  Variability (units) | 0.04 (0.02) | 0.04 (0.01) | 0.04 (0.01)
  Perseverations (units) | 0.06 (0.2) | 0.05 (0.2) | 0.04 (0.1)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Variability ANOVA; Test type: Superiority or Other; p = 0.397, ANOVA
Statistical Analysis 2: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; Perseverations ANOVA; Test type: Superiority or Other; p = 0.745, ANOVA
Statistical Analysis 3: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; 10mg vs 20mg variability; Test type: Superiority or Other; p = 0.362, t-test, 2 sided
Statistical Analysis 4: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; 10mg vs 20mg perseverations; Test type: Superiority or Other; p = 0.745, t-test, 2 sided

19. Post Hoc Outcome: Hit Reaction Time (Double Blind)
Description: Hit reaction time represents the average number of milliseconds required for a participant to respond to target stimuli. There are no meaningful absolute minimum or maximum scores, though 101ms is the current fastest verified response time per our review. A higher score is WORSE.
  This was not a pre-specified variable or an intentional post-hoc analysis, but it is calculated automatically and included here only for completeness of data submission.
Time Frame: Visits 2 vs 3 vs 4 on randomized medication doses.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Participants With Epilepsy: Placebo | Participants With Epilepsy: Methylphenidate 10 mg Dose | Participants With Epilepsy: Methylphenidate 20 mg
Number analyzed (Participants) | 31 | 31 | 31
ms | 437.4 (68.9) | 433.9 (65.2) | 435.6 (68.9)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Placebo vs Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; HRT ANOVA; Test type: Superiority or Other; p = 0.48, ANOVA
Statistical Analysis 2: Comparison: Participants With Epilepsy: Methylphenidate 10 mg Dose vs Participants With Epilepsy: Methylphenidate 20 mg; HRT 10mg vs 20mg; Test type: Superiority or Other; p = 0.793, t-test, 2 sided

20. Post Hoc Outcome: Hit Reaction Time (Open-Label)
Description: as for outcome 19
Time Frame: Visits 2 vs 3 vs 4 on randomized medication doses.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Participants With Epilepsy: Visit 1 (Baseline) | Participants With Epilepsy: Visit 5 (Open Label) | Healthy Controls: Visit 1 (Baseline) | Healthy Controls: Visit 5
Number analyzed (Participants) | 28 | 28 | 14 | 14
Milliseconds | 431.2 (69.4) | 425.7 (60.2) | 447.7 (62.2) | 423.4 (63.3)
Statistical Analysis 1: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label); HRT v1 vs v5 epilepsy; Test type: Superiority or Other; p = 0.5, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; HRT v1 vs v5 healthy; Test type: Superiority or Other; p = 0.075, t-test, 2 sided
Statistical Analysis 3: Comparison: Participants With Epilepsy: Visit 1 (Baseline) vs Participants With Epilepsy: Visit 5 (Open Label) vs Healthy Controls: Visit 1 (Baseline) vs Healthy Controls: Visit 5; HRT epilepsy vs healthy ANOVA; Test type: Superiority or Other; p = 0.2, ANOVA

ADVERSE EVENTS:
Time Frame: During entirety of pt participation (~2 months), throughout entirety of study.
Description: Commonly-expected side effects (anxiety, tachycardia) were routinely asked about at the end of participant visits, and responses recorded. Vital signs were checked at visits 1, 4, and 5. Fatigue was reported spontaneously by the affected participant and was not assessed routinely.
Groups:
- Placebo, 20mg, Then 10mg (Double-blind): Participants will receive three single doses of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and will complete cognitive testing and neuropsychiatric questionnaires. This single-dose phase will be followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy will first receive blinded, single-dose capsules in the following order:
  Placebo, 20mg of methylphenidate, 10mg of methylphenidate.
  At each visit, they will receive one capsule and then complete the neurocognitive batteries and neuropsychiatric questionnaires. There will be no medication administered between visits during this time. Following the final randomized visit, interested participants will be prescribed 10mg of methylphenidate twice daily, to be increased to 20mg of methylphenidate twice daily. After four weeks, their scores on the batteries and questionnaires will again be assessed.
- Placebo, 10mg, Then 20mg (Double-blind): Participants will receive three single doses of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and will complete cognitive testing and neuropsychiatric questionnaires. This single-dose phase will be followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy will first receive blinded, single-dose capsules in the following order:
  Placebo, 10mg of methylphenidate, 20mg of methylphenidate.
  At each visit, they will receive one capsule and then complete the neurocognitive batteries and neuropsychiatric questionnaires. There will be no medication administered between visits during this time. Following the final randomized visit, interested participants will be prescribed 10mg of methylphenidate twice daily, to be increased to 20mg of methylphenidate twice daily. After four weeks, their scores on the batteries and questionnaires will again be assessed.
- 10mg, 20mg, Then Placebo (Double-blind): Participants will receive three single doses of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and will complete cognitive testing and neuropsychiatric questionnaires. This single-dose phase will be followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy will first receive blinded, single-dose capsules in the following order:
  10mg of methylphenidate, 20mg of methylphenidate, Placebo.
  At each visit, they will receive one capsule and then complete the neurocognitive batteries and neuropsychiatric questionnaires. There will be no medication administered between visits during this time. Following the final randomized visit, interested participants will be prescribed 10mg of methylphenidate twice daily, to be increased to 20mg of methylphenidate twice daily. After four weeks, their scores on the batteries and questionnaires will again be assessed.
- 10mg, Placebo, Then 20mg (Double-blind): Participants will receive three single doses of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and will complete cognitive testing and neuropsychiatric questionnaires. This single-dose phase will be followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy will first receive blinded, single-dose capsules in the following order:
  10mg of methylphenidate, Placebo, 20mg of methylphenidate.
  At each visit, they will receive one capsule and then complete the neurocognitive batteries and neuropsychiatric questionnaires. There will be no medication administered between visits during this time. Following the final randomized visit, interested participants will be prescribed 10mg of methylphenidate twice daily, to be increased to 20mg of methylphenidate twice daily. After four weeks, their scores on the batteries and questionnaires will again be assessed.
- 20mg, 10mg, Then Placebo (Double-blind): Participants will receive three single doses of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and will complete cognitive testing and neuropsychiatric questionnaires. This single-dose phase will be followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy will first receive blinded, single-dose capsules in the following order:
  20mg of methylphenidate, 10mg of methylphenidate, Placebo.
  At each visit, they will receive one capsule and then complete the neurocognitive batteries and neuropsychiatric questionnaires. There will be no medication administered between visits during this time. Following the final randomized visit, interested participants will be prescribed 10mg of methylphenidate twice daily, to be increased to 20mg of methylphenidate twice daily. After four weeks, their scores on the batteries and questionnaires will again be assessed.
- 20mg, Placebo, Then 10mg (Double-blind): Participants will receive three single doses of blinded medication, either a placebo, 20mg of methylphenidate, or 10mg of methylphenidate, and will complete cognitive testing and neuropsychiatric questionnaires. This single-dose phase will be followed by an open-label 4-week treatment trial of methylphenidate.
  Methylphenidate: Participants with epilepsy will first receive blinded, single-dose capsules in the following order:
  20mg of methylphenidate, Placebo, 10mg of methylphenidate.
  At each visit, they will receive one capsule and then complete the neurocognitive batteries and neuropsychiatric questionnaires. There will be no medication administered between visits during this time. Following the final randomized visit, interested participants will be prescribed 10mg of methylphenidate twice daily, to be increased to 20mg of methylphenidate twice daily. After four weeks, their scores on the batteries and questionnaires will again be assessed.
- Healthy Controls: Healthy controls will complete the same neurocognitive batteries and neuropsychiatric questionnaires as individuals with epilepsy, but will not be exposed to study medication. They are included as a control group for the open-label phase of the study (visit 1 vs visit 5) only.
Arm/Group | Participants With Epilepsy (Open-label) | Placebo, 20mg, Then 10mg (Double-blind) | Placebo, 10mg, Then 20mg (Double-blind) | 10mg, 20mg, Then Placebo (Double-blind) | 10mg, Placebo, Then 20mg (Double-blind) | 20mg, 10mg, Then Placebo (Double-blind) | 20mg, Placebo, Then 10mg (Double-blind) | 40mg, 20mg, Then Placebo (One Participant) | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/5 | 0/1 | 0/15
Other Adverse Events (participants affected / at risk) | 2/30 | 0/6 | 1/6 | 0/5 | 1/6 | 2/6 | 0/5 | 1/1 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Epilepsy (Open-label) (N=30) | Placebo, 20mg, Then 10mg (Double-blind) (N=6) | Placebo, 10mg, Then 20mg (Double-blind) (N=6) | 10mg, 20mg, Then Placebo (Double-blind) (N=5) | 10mg, Placebo, Then 20mg (Double-blind) (N=6) | 20mg, 10mg, Then Placebo (Double-blind) (N=6) | 20mg, Placebo, Then 10mg (Double-blind) (N=5) | 40mg, 20mg, Then Placebo (One Participant) (N=1) | Healthy Controls (N=15)
Anxiety/panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Four participants experienced a period of anxiety following ingestion of medication, lasting 1-3 hours, without other symptoms. Vitals were stable, and symptoms resolved on their own. Two of the four elected to withdraw.
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — ~4 hours after dose had 2-3 hours of HR ~160bpm w/ no other symptoms. Resolved w/ no intervention. No other symptoms. BP stable per pt report. Pt did not seek care. We withdrew pt.
Increased anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — One participant reported increased anxiety after having tolerated all of the blinded capsules in the randomized portion. This participant elected to withdraw from the open- label portion.
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — One participant tolerated all three randomized doses, yet experienced fatigue on the open-label dose. This participant elected to withdraw from the open-label trial.

LIMITATIONS AND CAVEATS:
Relatively small sample; Control is healthy patients rather than epilepsy patients; Healthy controls improve more on re-testing than epilepsy patients; Single-dose portion does not mirror clinical practice; open-label portion is not blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes